CLINICAL TRIAL: NCT04910139
Title: A User Study of the Soniflow System for Nasal Congestion Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Wave Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-001
Record Dates: First submitted 2021-05-23; First posted 2021-06-02 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment using acoustic energy
  Interventions: Device: Soniflow System

INTERVENTIONS:
Device: Soniflow System — Treatment using acoustic vibrational headband worn circumferentially at the level of the forehead paired with a Smartphone App.
  Other Names: Soniflow System to provide nasal congestion relief

SUMMARY:
The Soniflow System consists of an acoustic vibrational headband paired with a Smartphone App to provide rapid relief of nasal congestion.

DETAILED DESCRIPTION:
The Soniflow System is a non-invasive device to provide rapid relief of nasal congestion. It consists of a headband with ultrasound transducers (hardware) coupled to a Smartphone application (software).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >18 years of age
2. Subject has had moderate to severe symptoms of nasal congestion for >3 months (TNSS rating of 2 or 3)
3. Subject has signed IRB-approved informed consent form

Exclusion Criteria:

1. Subject has neurologic comorbidities
2. Subject has active dental infection
3. Subject is pregnant
4. Subject has implanted intracranial electrostimulation device(s) (e.g. cochlear implant, deep brain stimulator)
5. Subject has undergone sinonasal or craniomaxillofacial surgery within the lats 3 months
6. Subject has been diagnosed with intracranial hemorrhage within the last 6 months
7. Subject has open scalp wounds or rashes
8. Subject has any history of craniotomy without replacement of a bone flap
9. Subject has elevated sensitivity to sound
10. Any physical condition that in the investigator's opinion would prevent adequate study participation or pose increased risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Johnson, MD, Principal Investigator — Principal Investigator
Locations (1):
- San Francisco Otolaryngology Medical Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult subjects with nasal congestion
Arm/Group | Treatment
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0
  Age: Between 18 and 65 years | 46
  Age: >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50
Total Nasal Symptom Score [Mean (Inter-Quartile Range); unit: units on a scale] | 4.1 [3.5 to 4.6]

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Score
Description: TNSS is a measure of nasal congestion, measured as the sum of four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing (using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe). The minimum TNSS value is 0. The maximum TNSS value is 12. Lower TNSS score means a better outcome
Time Frame: 20 minutes
Population: Adult subjects with nasal congestion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 50
score on a scale | 2.0 [1.6 to 2.5]

2. Secondary Outcome: Visual Analog Scale (VAS) for Headache
Description: Visual Analog Scale (VAS) for Headache, using a scale of 0-10. 0 is the minimum and 10 is maximum on this scale. Lower scores mean a better outcome.
Time Frame: 20 minutes
Population: adults with nasal congestion
Measure: Mean (95% Confidence Interval); unit: score on a scale of 0-10
Arm/Group | Treatment
Number analyzed (Participants) | 50
score on a scale of 0-10 | 0.9 [0.4 to 1.5]

3. Secondary Outcome: Visual Analog Scale (VAS) for Facial Pain
Description: Visual Analog Scale (VAS) for Facial Pain, using a scale of 0-10. 0 is minimum and 10 is the maximum value for this scale. Lower scores mean a better outcome.
Time Frame: 20 minutes
Population: adults with nasal congestion
Measure: Mean (95% Confidence Interval); unit: score on a scale (of 0-10)
Arm/Group | Treatment
Number analyzed (Participants) | 50
score on a scale (of 0-10) | 0.9 [0.5 to 1.5]

ADVERSE EVENTS:
Time Frame: 1 day, acute study
Description: Adverse event definition is same as clinicaltrials.gov definition. Adverse events were collected for all 50 participants
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04910139/Prot_SAP_001.pdf